CLINICAL TRIAL: NCT02153099
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Safety, Tolerability and Pharmacokinetic Study of Escalating Single Doses of ENV8058 in Healthy Subjects
Brief Title: Safety, Tolerability and Pharmacokinetics of Escalating Single Doses of ENV8058 (TAK-058) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ENV8058_101; U1111-1154-9569 (Other: World Health Organization)
Record Dates: First submitted 2014-05-29; First posted 2014-06-02 (Estimated); Results first posted 2015-12-17 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-11

CONDITIONS: Dose Finding Study
Keywords: Drug therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- Cohort 1: TAK-058 15 mg (Experimental): TAK-058 15 mg, 100 mL oral solution, once on Day 1.
  Interventions: Drug: TAK-058 (ENV8058)
- Cohort 2: TAK-058 30 mg (Experimental): TAK-058 30 mg, 100 mL oral solution, once on Day 1.
  Interventions: Drug: TAK-058 (ENV8058)
- Cohort 3: TAK-058 45 mg (Experimental): TAK-058 45 mg, 100 mL oral solution, once on Day 1.
  Interventions: Drug: TAK-058 (ENV8058)
- Cohort 4: TAK-058 5 mg (Experimental): TAK-058 5 mg, 100 mL oral solution, once on Day 1.
  Interventions: Drug: TAK-058 (ENV8058)
- Cohort 5: TAK-058 75 mg (Experimental): TAK-058 75 mg, 100 mL oral solution, once on Day 1.
  Interventions: Drug: TAK-058 (ENV8058)
- Cohort 6: TAK-058 150 mg (Experimental): TAK-058 150 mg, 100 mL oral solution, once on Day 1.
  Interventions: Drug: TAK-058 (ENV8058)
- Cohort 1-6: Placebo (Placebo Comparator): TAK-058 placebo-matching, 100 mL oral solution, once on Day 1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TAK-058 (ENV8058) — TAK-058 (ENV8058) oral solution
  Arms: Cohort 1: TAK-058 15 mg; Cohort 2: TAK-058 30 mg; Cohort 3: TAK-058 45 mg; Cohort 4: TAK-058 5 mg; Cohort 5: TAK-058 75 mg; Cohort 6: TAK-058 150 mg
Drug: Placebo — TAK-058 (ENV8058) placebo-matching oral solution
  Arms: Cohort 1-6: Placebo

SUMMARY:
The purpose of this study is to characterize the safety and tolerability profile of escalating dose levels of ENV8058 (TAK-058) solution when administered as a single oral dose in healthy adults.

DETAILED DESCRIPTION:
The drug being tested in this study is called ENV8058 (also known as TAK-058). ENV8058 is being tested to find a safe and well-tolerated dose and to assess how ENV8058 moves throughout the body. This study will look at side effects and lab results in people who took ENV8058. This study was designed as a randomized, sequential-panel, single rising dose study.

The study population will consist of 6 Cohorts with 8 participants in each Cohort; with 6 participants randomized to receive a single dose of ENV8058, and 2 participants to receive placebo. Participants in each Cohort will receive a single dose of study drug after a 10-hour fast. The starting dose is 15 mg followed by administrations of 30, 45, 15, 75 and 150 mg.

* ENV8058 (Tak-058): 5, 15, 30, 45, 75 or 150 mg oral solution
* Placebo (dummy inactive) - this oral solution looks like the study drug but has no active ingredient

This single-centre trial will be conducted in the United States. The overall time to participate in this study is up to 14 days. Participants will make 2 visits to the clinic, including one 5-day period of confinement to the clinic. All participants will be contacted by telephone 14 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures including requesting that a participant fast for any laboratory evaluations.
3. Is a healthy male or female adult who is 18 to 55 years of age inclusive at the time of informed consent and study drug dosing.
4. Weighs at least 45 kg (99 lbs) and has a body mass index (BMI) between 18.0 and 30.0 kg/m^2, inclusive at Screening.
5. A male participant who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent throughout the duration of the study and for 12 weeks after last dose.
6. A female participant with no childbearing potential, defined as the participant has been surgically sterilized (hysterectomy, bilateral oophorectomy or tubal ligation) or who are postmenopausal (defined as continuous amenorrhea of at least 2 years and follicle-stimulating hormone (FSH)>40 IU/L).

Exclusion Criteria:

1. Has received any investigational compound within 30 days prior to the first dose of study medication.
2. Is an immediate family member, study site employee, or is in a dependant relationship with a study site employee who is involved in the conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
3. Has uncontrolled, clinically significant neurologic, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, urologic, immunologic, endocrine disease, or psychiatric disorder, or other abnormality, which may impact the ability of the participant to participate or potentially confound the study results.
4. Has a known hypersensitivity to any component of the formulation of ENV8058 (TAK-058).
5. Has a positive urine drug result for drugs of abuse at Screening or Check-in (Day -1).
6. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 1 year prior to the Screening Visit or is unwilling to agree to abstain from alcohol and drugs throughout the study.
7. Has taken any excluded medication, supplements, or food products listed in the Excluded Medications and Dietary Products table.
8. If female, the participant is of childbearing potential (e.g premenopausal, not sterilized).
9. If male, the participant intends to donate sperm during the course of this study or for 12 weeks thereafter.
10. Has evidence of current cardiovascular, central nervous system, hepatic, hematopoietic disease, renal dysfunction, metabolic or endocrine dysfunction, serious allergy, asthma hypoxemia, hypertension, seizures, or allergic skin rash. There is any finding in the participant's medical history, physical examination, or safety laboratory tests giving reasonable suspicion of a disease that would contraindicate taking ENV8058 (TAK-058), or a similar drug in the same class, or that might interfere with the conduct of the study. This includes, but is not limited to seizure disorders and cardiac arrhythmias.
11. Has previously had a seizure or convulsion (lifetime), including absence seizure and febrile convulsion.
12. Has current or recent (within 6 months) gastrointestinal disease that would be expected to influence the absorption of drugs (ie, a history of malabsorption, any surgical intervention known to impact absorption [eg, bariatric surgery or bowel resection], esophageal reflux, peptic ulcer disease, erosive esophagitis, or frequent [more than once per week] occurrence of heartburn).
13. Has a history of cancer or other malignancy, except basal cell carcinoma that has been in remission for at least 5 years prior to Day 1.
14. Has a positive test result for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody or a known history of human immunodeficiency virus infection at Screening.
15. Has used nicotine-containing products (including but not limited to cigarettes, electronic cigarettes, pipes, cigars, chewing tobacco, nicotine patch or nicotine gum) within 28 days prior to Check-in (Day -1). Cotinine test is positive at Screening or Check-in (Day -1).
16. Has poor peripheral venous access.
17. Has donated or lost 450 mL or more of his or her blood volume (including plasmapheresis), or had a transfusion of any blood product within 45 days prior to Day 1.
18. Has a Screening or Check-in (Day -1) abnormal (clinically significant) electrocardiogram (ECG). Entry of any participant with an abnormal (not clinically significant) ECG must be approved and documented by signature by the principal investigator or medically qualified subinvestigator.
19. Subject had a supine blood pressure outside the ranges of 90 to 140 mm Hg for systolic and 60 to 90 mm Hg (males) and 50 to 90 mm Hg (females) for diastolic, confirmed with 1repeat testing, at the Screening Visit or Check-in (Day -1).
20. Has a resting heart rate outside the range 40 to 90 bpm, confirmed with one repeat testing, at the Screening Visit or Check-in (Day -1).
21. Has a QT interval with Fridericia's correction method (QTcF) >430 ms (males) or >450 ms (females) or PR outside the range of 120 to 220 ms, confirmed with one repeat testing, at the Screening Visit or Check-in (Day -1) Visit.
22. Has abnormal Screening or Check-in (Day -1) laboratory values that suggest a clinically significant underlying disease or participant with the following lab abnormalities: alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >1.5 the upper limits of normal.
23. Has a risk of suicide according to the Investigator's clinical judgment (eg, per Columbia-Suicide Severity Rating Scale [CSSRS] or has made a suicide attempt in the previous 6 months.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2014-06; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (1):
- Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 14 May 2014 (signing of informed consent) to 13 November 2014.
Pre-assignment Details: Healthy Volunteers were enrolled in 1 of 6 Dose Cohorts: (5 mg, 15 mg, 30 mg, 45 mg, 75 mg, 150 mg TAK-058) or placebo.
Groups:
- Cohort 4: TAK-058 5 mg: TAK-058 (ENV8058) 5 mg, 100 mL oral solution, once on Day 1.
- Cohorts 6: TAK-058 150 mg: TAK-058 150 mg, 100 mL oral solution, once on Day 1.
Period: Overall Study
Arm/Group | Cohort 4: TAK-058 5 mg | Cohort 1: TAK-058 15 mg | Cohort 2: TAK-058 30 mg | Cohort 3: TAK-058 45 mg | Cohort 5: TAK-058 75 mg | Cohorts 6: TAK-058 150 mg | Cohort 1-6: Placebo
Started | 6 | 6 | 6 | 6 | 6 | 6 | 12
Completed | 6 | 6 | 6 | 6 | 6 | 6 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 4: TAK-058 5 mg | Cohort 1: TAK-058 15 mg | Cohort 2: TAK-058 30 mg | Cohort 3: TAK-058 45 mg | Cohort 5: TAK-058 75 mg | Cohorts 6: TAK-058 150 mg | Cohort 1-6: Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.7 (11.38) | 37.0 (14.01) | 35.3 (10.71) | 34.2 (7.78) | 41.5 (10.93) | 30.8 (8.54) | 34.2 (9.11) | 35.1 (10.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 2 | 1 | 0 | 2 | 9
  Male | 5 | 5 | 4 | 4 | 5 | 6 | 10 | 39
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 3
  Black or African American | 2 | 1 | 1 | 1 | 3 | 1 | 3 | 12
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  White | 3 | 5 | 5 | 4 | 3 | 5 | 7 | 32
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 0 | 3 | 1 | 3 | 1 | 2 | 2 | 12
  Non-Hispanic or non-Latino | 6 | 3 | 5 | 3 | 5 | 4 | 10 | 36
Region of Enrollment [Number; unit: participants]
  North America | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 48
Height [Mean (Standard Deviation); unit: cm] | 171.2 (4.40) | 167.7 (6.44) | 174.7 (15.20) | 170.2 (10.42) | 178.7 (8.78) | 175.5 (8.69) | 176.1 (12.91) | 173.8 (10.49)
Weight [Mean (Standard Deviation); unit: kg] | 72.73 (10.683) | 70.65 (6.763) | 81.72 (20.142) | 79.38 (10.860) | 86.17 (12.796) | 80.50 (16.471) | 72.77 (12.359) | 77.09 (13.514)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 24.79 (3.110) | 25.11 (1.674) | 26.35 (3.086) | 27.39 (2.440) | 26.86 (1.989) | 25.89 (2.728) | 23.42 (2.533) | 25.40 (2.770)
Smoking Status [Number; unit: participants]
  Never smoked | 5 | 5 | 5 | 6 | 5 | 5 | 11 | 42
  Current smoker | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Ex-smoker | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 6
Caffeine Consumption [Number; unit: participants]
  Yes | 3 | 3 | 4 | 4 | 4 | 3 | 6 | 27
  No | 3 | 3 | 2 | 2 | 2 | 3 | 6 | 21
Female Reproductive Status [Number; unit: participants]
  Postmenopausal | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 3
  Surgically Sterile | 0 | 0 | 1 | 2 | 1 | 0 | 2 | 6
  Female of Childbearing Potential | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Subject is Male | 5 | 5 | 4 | 4 | 5 | 6 | 10 | 39

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experience at Least One Treatment Emergent Adverse Event (TEAE)
Description: Treatment-emergent adverse events are defined as any unfavorable and unintended sign, symptom or disease temporally associated with the use of a medicinal product reported from first dose of study drug through 14 days after the last dose of study drug, or if a serious adverse event, within 30 days after the last dose of study drug.
Time Frame: Baseline up to Day 30
Population: Safety population included all enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 4: TAK-058 5 mg | Cohort 1: TAK-058 15 mg | Cohort 2: TAK-058 30 mg | Cohort 3: TAK-058 45 mg | Cohort 5: TAK-058 75 mg | Cohorts 6: TAK-058 150 mg | Cohort 1-6: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12
percentage of participants | 16.7 | 0 | 50.0 | 0 | 16.7 | 0 | 8.3

2. Primary Outcome: Percentage of Participants With Markedly Abnormal Safety Laboratory Tests
Description: The percentage of participants with any markedly abnormal standard safety laboratory values, including hematology, serum chemistries, and urinalysis, during the treatment period.
Time Frame: Baseline up to Day 14
Population: Safety population included all enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 4: TAK-058 5 mg | Cohort 1: TAK-058 15 mg | Cohort 2: TAK-058 30 mg | Cohort 3: TAK-058 45 mg | Cohort 5: TAK-058 75 mg | Cohorts 6: TAK-058 150 mg | Cohort 1-6: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12
percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Percentage of Participants With Markedly Abnormal Vital Sign Measurements
Description: The percentage of participants who meet markedly abnormal criteria for vital signs, including oral body temperature, respiration rate, pulse [beats per minute (bpm)], and resting blood pressure and after standing.
Time Frame: Baseline up to Day 14
Population: Safety population included all enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 4: TAK-058 5 mg | Cohort 1: TAK-058 15 mg | Cohort 2: TAK-058 30 mg | Cohort 3: TAK-058 45 mg | Cohort 5: TAK-058 75 mg | Cohorts 6: TAK-058 150 mg | Cohort 1-6: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12
percentage of participants
  Any Vital Sign - Abnormal Low | 66.7 | 16.7 | 33.3 | 33.3 | 50.0 | 16.7 | 50.0
  Any Vital Sign - Abnormal High | 0 | 16.7 | 0 | 0 | 0 | 16.7 | 0
  Any Vital Sign - Any Abnormality | 66.7 | 33.3 | 33.3 | 33.3 | 50.0 | 33.3 | 50.0
  Systolic Blood Pressure <85 mmHg | 16.7 | 0 | 33.3 | 0 | 0 | 16.7 | 0
  Systolic Blood Pressure >180 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Systolic Blood Pressure - Any Abnormality | 16.7 | 0 | 33.3 | 0 | 0 | 16.7 | 0
  Diastolic Blood Pressure <50 mmHg | 0 | 0 | 0 | 16.7 | 16.7 | 0 | 0
  Diastolic Blood Pressure >110 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Diastolic Blood Pressure - Any Abnormality | 0 | 0 | 0 | 16.7 | 16.7 | 0 | 0
  Pulse <50 bpm | 50.0 | 16.7 | 16.7 | 16.7 | 50.0 | 0 | 33.3
  Pulse >120 bpm | 0 | 16.7 | 0 | 0 | 0 | 16.7 | 0
  Pulse - Any Abnormality | 50.0 | 33.3 | 16.7 | 16.7 | 50.0 | 16.7 | 33.3
  Temperature <35.6 degrees Celsius | 16.7 | 0 | 0 | 0 | 0 | 0 | 25.0
  Temperature >37.7 degrees Celsius | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Temperature - Any Abnormality | 16.7 | 0 | 0 | 0 | 0 | 0 | 25.0

4. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for ENV8058 (TAK-058)
Description: Maximum observed plasma concentration (Cmax) is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve.
Time Frame: Predose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, and 96 hours postdose
Population: Pharmacokinetic (PK) Population included all enrolled participants.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 4: TAK-058 5 mg | Cohort 1: TAK-058 15 mg | Cohort 2: TAK-058 30 mg | Cohort 3: TAK-058 45 mg | Cohort 5: TAK-058 75 mg | Cohorts 6: TAK-058 150 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
ng/mL | 142.4 (43.68) | 565.0 (112.07) | 824.7 (297.45) | 1248.2 (254.06) | 1563.3 (339.51) | 2136.7 (818.04)

5. Secondary Outcome: AUC(0-tlqc): Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for ENV8058 (TAK-058)
Description: (AUC(0-tlqc) is a measure of total plasma exposure to the drug from time 0 to time of the last quantifiable concentration (AUC[0-tlqc]).
Time Frame: Predose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, and 96 hours postdose
Population: PK Population included all enrolled participants.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Cohort 4: TAK-058 5 mg | Cohort 1: TAK-058 15 mg | Cohort 2: TAK-058 30 mg | Cohort 3: TAK-058 45 mg | Cohort 5: TAK-058 75 mg | Cohorts 6: TAK-058 150 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
ng*hr/mL | 617.8 (334.31) | 2297.8 (678.69) | 3243.9 (1261.96) | 5027.3 (1001.82) | 6275.4 (1535.27) | 9385.8 (3398.36)

6. Secondary Outcome: AUC(0-inf): Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for ENV8058 (TAK-058)
Description: AUC(0-inf) is a measure of total plasma exposure to the drug from time zero extrapolated to infinity.
Time Frame: Predose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, and 96 hours postdose
Population: PK Population included all enrolled participants.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Cohort 4: TAK-058 5 mg | Cohort 1: TAK-058 15 mg | Cohort 2: TAK-058 30 mg | Cohort 3: TAK-058 45 mg | Cohort 5: TAK-058 75 mg | Cohorts 6: TAK-058 150 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
ng*hr/mL | 620.5 (334.86) | 2305.5 (678.59) | 3252.1 (1264.03) | 5038.9 (998.48) | 6292.1 (1546.90) | 9407.9 (3402.50)

7. Secondary Outcome: Terminal Elimination Half-life (T1/2) Pharmacokinetic Parameter for ENV8058 (TAK-058)
Description: Terminal Phase Elimination Half-life (T1/2) is the time required for half of the drug to be eliminated from the plasma.
Time Frame: Predose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, and 96 hours postdose
Population: PK population included all enrolled participants.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort 4: TAK-058 5 mg | Cohort 1: TAK-058 15 mg | Cohort 2: TAK-058 30 mg | Cohort 3: TAK-058 45 mg | Cohort 5: TAK-058 75 mg | Cohorts 6: TAK-058 150 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
hours | 2.814 (1.0871) | 5.300 (2.2727) | 5.925 (4.5780) | 9.611 (7.3329) | 10.486 (7.1865) | 8.601 (7.9332)

ADVERSE EVENTS:
Time Frame: First dose of study drug to 14 days after the last dose of study drug, or if a serious adverse event, within 30 days after the last dose of study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Cohort 4: TAK-058 5 mg | Cohort 1: TAK-058 15 mg | Cohort 2: TAK-058 30 mg | Cohort 3: TAK-058 45 mg | Cohort 5: TAK-058 75 mg | Cohorts 6: TAK-058 150 mg | Cohort 1-6: Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/12
Other Adverse Events (participants affected / at risk) | 1/6 | 0/6 | 3/6 | 0/6 | 1/6 | 0/6 | 1/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 4: TAK-058 5 mg (N=6) | Cohort 1: TAK-058 15 mg (N=6) | Cohort 2: TAK-058 30 mg (N=6) | Cohort 3: TAK-058 45 mg (N=6) | Cohort 5: TAK-058 75 mg (N=6) | Cohorts 6: TAK-058 150 mg (N=6) | Cohort 1-6: Placebo (N=12)
Infrequent bowel movements (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Euphoric mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.